CLINICAL TRIAL: NCT02163473
Title: Hypoxia Inducible Factor 1 Alpha as a Novel Biomarker in Septic Shock
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201200142
Record Dates: First submitted 2014-06-05; First posted 2014-06-13 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Septic patients: Blood Draw Biological samples: The investigators will collect blood and compare the expression of HIF complex in 3 distinct ways: between patients and controls, within the same patient in a time-dependent fashion, and between different patients.
  Interventions: Procedure: Septic patients
- Healthy Control: The investigators will collect blood and compare the expression of HIF complex in 3 distinct ways: between patients and controls, within the same patient in a time-dependent fashion, and between different patients.
  Interventions: Procedure: Healthy Control

INTERVENTIONS:
Procedure: Septic patients — The investigators will draw two sets of blood samples. One at baseline, 10 mL, and another, 24 hours later, 10 mL, for a total of 20 mL.
  Groups: Septic patients
Procedure: Healthy Control — The investigators will draw 10 mL, once, during baseline for a total of 10 mL among the healthy control group.
  Groups: Healthy Control

SUMMARY:
The purpose of this research study is to determine if a chemical marker in the blood, hypoxia-inducible factor (HIF-1 alpha), can be used to predict subject's hospital outcomes when the subject is diagnosed with sepsis. Sepsis is defined as either the presence of pathogenic organisms or their toxins in the blood and tissues. Sepsis is one of the most significant challenges in critical care medicine. The investigators propose that hypoxia-induced expression of HIF-1 alpha will correlate with the clinical features of Sepsis and in the future, HIF-1 alpha may be used as a biomarker in Sepsis.

DETAILED DESCRIPTION:
Sepsis is one of the most significant challenges in critical care. Septic shock (SS) is the most severe form of sepsis and is associated with higher mortality, significant financial expenses and longer lengths of stay. Pathophysiological mechanisms of SS include 3 key components: 1) bacterial overgrowth, 2) spill of bacterial product into the blood causing hemodynamic insufficiency, and 3) both lead to tissue hypoxia (TH). To date the biomarkers of sepsis/SS are limited to hemodynamic parameters. However, aggressive fluid resuscitation does not fully prevent development of tissue hypoxia (TH). To date the investigators are limited in appreciating TH by measurement of lactic acid (LA), which is neither an early nor an accurate marker. Unfortunately, LA has limited predictive value in SS due to its complex metabolism. Thus, there is an acute need for biomarkers that would aid diagnosis and prognosis of sepsis/septic shock.

Cellular responses/adaptations to hypoxia rely on the transcription hypoxia-inducible factor HIF, a heterodimeric protein composed of a constitutively expressed subunit and an inducible (types 1, 2, and 3) subunit. More recently HIF was identified in diverse tissues including blood; it has been also shown that HIF expression in blood cells is representative of systemic tissues in hypoxic conditions.

ELIGIBILITY:
Inclusion Criteria: Septic patients

* Age 18 ≤ 80 years
* Negative pregnancy test for women of childbearing potential
* Meets two or more of Systemic Inflammatory Response System (SIRS) criteria (tachypnea, tachycardia, hypo/hyperthermia, leukopenia/leukocytosis)
* Evidence of tissue hypo-perfusion, or organ dysfunction by any of the following
* Sepsis induced hypotension with systolic blood pressure <90
* Lactate above 1.5 mmol/Liter
* Urine output below 0.5 mL/kg/hr for more than 2 hours despite adequate fluid resuscitation
* Tissue hypoxia
* Bilirubin > 2 mg/dl in absence of liver cirrhosis
* Creatinine (CR)> 2.0 mg/dL, Acute Kidney Injury as evident by CR increase by 0.5 mg/dL from baseline
* Platelet count < 100,000
* Coagulopathy with international normalized ratio (INR) >1.5

Inclusion: Healthy Controls

* Age and gender-matched to sepsis patients
* Negative pregnancy test in women of childbearing potential
* Never smoker (<1 pack year history)

Exclusion Criteria: Septic patients

* History of Malignancy, including carcinoma during the preceding 5 years.
* Recent surgery, within 48 hours, or anticipated surgery within 24 hours
* Contraindication for neck/chest central venous line
* History of cardiopulmonary resuscitation (CPR) prior to inclusion
* Transfer from another institution
* History of cirrhosis
* Transplant recipient
* Known HIV
* Use of ≥ 15 mg prednisone daily or equivalent
* Severe anemia: hematocrit ≤ 20

Exclusion: Healthy Controls

* History of Malignancy, including carcinoma during the preceding 5 years.
* Taking any prescription medications, other than any type of prescribed hormonal birth control.
* Current smoking history and/or > 1 pack year history
* Current use (within the last week) anti-inflammatory medications, such as aspirin, ibuprofen, naproxen and/or prednisone

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal healthy controls recruited from the community. Subjects with sepsis admitted to the University of Florida Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Hypoxia-inducible factor as a predictive biomarker of sepsis. | Baseline,
  Hypoxia-inducible factor will be measured at initial diagnosis (baseline) and 24 hours later in subjects with clinical presentation of sepsis and correlated with lactic acidosis.
Hypoxia-inducible factor as a predictive biomarker of sepsis | 24 hours
  Hypoxia-inducible factor will be measured at initial diagnosis (baseline) and 24 hours later in subjects with clinical presentation of sepsis and correlated with lactic acidosis.

SECONDARY OUTCOMES:
Evaluate the role of HIF complex as biomarker and its correlation with "Survive the Sepsis Campaign 2012" gold standard septic shock severity and morbidity/mortality predictors. | 28 days
  At discharge a detailed chart analysis will be performed for the first 24 hrs, survival at 28 day; correlations of clinical course-derived data and serum cytokine content with the HIF content/expression and function will be analyzed by Spearman's rank correlation test.

CONTACTS AND LOCATIONS:
Overall Officials: Wael Nasser, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States